CLINICAL TRIAL: NCT02516943
Title: The Effects of Using Pathological- Based Guidelines for Arterial Blood Gas Analysis in Patients Aftercardiac Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Si 723/2557(EC4)
Record Dates: First submitted 2015-08-04; First posted 2015-08-06 (Estimated); Last update posted 2015-12-11 (Estimated); Status verified 2015-12

CONDITIONS: Blood Gas Analysis
Keywords: Arterial blood gas analysis
MeSH Terms: interventions — Guidelines as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Active Comparator): The patient were retrospectively included according to the last digit of their admission number (odd number). The had arterial blood gas analysis every 4 hour during the ICU stay.
  Interventions: Other: Control
- Guideline (Active Comparator): The patient were prospectively included and they had arterial blood gas analysis following the pathological- based guidelines for arterial blood gas analysis in patients aftercardiac surgery
  Interventions: Other: Guideline

INTERVENTIONS:
Other: Control — The patient's ABGs were test according to a 4 - hour routine
  Arms: Control
Other: Guideline — The patient's ABGs were test according to the guideline for requests Arterial Blood Gas status post cardiac surgery
  Arms: Guideline

SUMMARY:
Blood gas analysis were routinely monitor every 4 hours in our surgical cardiac intensive care unit (SICU). These luxury investigations waste the resources. Therefore we develop a pathological- based guideline for arterial blood gas analysis in patients after cardiac surgery. We test the guideline for its safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergone elective cardiac surgery with cardiopulmonary bypass

Exclusion Criteria:

* Emergency surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2014-11; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Number of ABG test | 14 days
  during intensive care stay

SECONDARY OUTCOMES:
Influence of ABG testing on patients' outcome. | 14 days
  during intensive care stay

CONTACTS AND LOCATIONS:
Overall Officials: Sirilak Suksompong, MD, Principal Investigator — Mahidol University